CLINICAL TRIAL: NCT03674983
Title: PrEP Seguro: Antiretroviral-based HIV Prevention Among Men at High Risk in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Consorcio de Investigación sobre VIH/SIDA/TB (CISIDAT). (Other); University of California, San Francisco (Other); Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Omar Galarraga, PhD, Associate Professor of Health Services, Policy and Practice, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R34MH114664-01 (NIH); 5R34MH114664-02 (NIH)
Record Dates: First submitted 2018-08-10; First posted 2018-09-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: adherence; AIDS prevention; Anti-Retroviral Agents; Behavioral Economics; Biological Markers; Cost-effectiveness; MSM; HIV Prevention; PrEP
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Aim 1: discrete choice experiment (DCE) with n=200. Aim 2: randomly assign 100 HIV-negative MSW in a 1:1 ratio either to: the SoC group, or to the CEI group. MSW in the SoC group (n=50) will receive transport reimbursement at baseline, 3 and 6 months. MSW in the CEI group (n=50) will receive transport reimbursement at baseline, 3 and 6 months, and additional incentives based on sufficiently high PrEP adherence at months 3 and 6. All participants will provide hair samples and have optional brief counseling based on hair sample results. Those in the CEI group, will receive additional incentives if concentrations of TDF/FTC in hair samples corroborate that they have been sufficiently adherent in recent weeks. The final incentives (amounts, format, location, etc.) will be based on Aim 1 results. 1-2 weeks after study visits, participants will receive a grade depending on the drug level detected in their scalp hair. The CEI amounts will be distributed depending on grade.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEI Group (Experimental): CEI Group will receive the standard of care (information, prescription, free PrEP) and economic incentives contingent on sufficiently-high adherence to PrEP.
  Interventions: Behavioral: Conditional Economic Incentive (CEI)
- SOC Group (No Intervention): SOC Group will receive the standard of care only (information, prescription, free PrEP.)

INTERVENTIONS:
Behavioral: Conditional Economic Incentive (CEI) — If hair testing shows that a participant has taken PrEP pills about 5-7 times in the previous week, he will receive a grade "A"; if he has taken PrEP pills about 3-4 times in the previous week he will receive a grade "B"; and if he has taken PrEP pills only 2 times or less, he will receive a grade "C". For those in the CEI group, if participant gets an A, he receives two additional prizes; if he gets a B, he receives one additional prize; and if he gets a C, he receives no additional prizes.
  Arms: CEI Group

SUMMARY:
The objective of this R34 application is to prepare for testing innovative user-centered ways to promote PrEP adherence at scale. Our central hypothesis is that adherence to PrEP can be improved among MSW if PrEP is provided for free along with highly-tailored conditional economic incentives (CEI). The specific aims are: Aim 1: To refine the design of PrEP adherence intervention with user-centered conditional economic incentives to maximize sustained adherence behaviors through a user-responsive computerized survey (n=200). We incorporate quantitatively identified preferences for CEIs through a user- responsive computerized survey. We use conjoint analysis to understand preferences for CEI intervention components and how CEIs should be integrated into an optimal combination package to be tested in Aim 2. Aim 2: Measure the extent to which a user-centered CEI intervention can help MSW increase their adherence to free PrEP in a randomized controlled pilot (n=100). Among MSW who accept to take free PrEP, and return at month 1 for a second pill bottle, we will randomize n=100 MSW to either: standard of care (SoC: information, prescription, free PrEP) or CEI (SoC + incentives contingent on sufficiently-high adherence to PrEP). We will assess the primary outcome (biomarker of adherence using scalp hair analysis) at months 3 and 6, as well as secondary outcomes: clinic attendance/retention, medication possession ratio, self-reported PrEP use, and sexual behavioral disinhibition (number of partners, condom use, incident STI). Aim 3: Estimate the preliminary cost-effectiveness of incentives for PrEP adherence to maximize future policy and practice relevance of this promising intervention strategy. Our working hypothesis is that conditional economic incentives for PrEP adherence will be cost-effective in terms of cost per fully- adherent month on PrEP, cost per HIV infection averted, and cost per disability-adjusted life year saved when compared to controls not receiving the conditional incentives. The expected outcome of this R34 is a demonstration that is feasible to implement user-centered CEIs in this context, as well as preliminary efficacy and cost-effectiveness data. The project will have positive impact because it is a critical step toward scaled-up implementation of PrEP in this highly-at-risk population of MSWs in Mexico, with implications for other concentrated epidemics among MSW worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth and self-identifies as male at the time of enrollment
* At least 18 years of age
* Has tested negative for HIV in the past month
* Demonstrates high risk of HIV acquisition defined as having had sex with penetration (oral or anal) with at least 8 male partners in past six months
* Has exchanged or accepted money, drugs or gifts in exchange for sex on at least 8 occasions in the past month
* Willing and capable of providing blood and scalp hair samples for assessments
* Willing and able to provide written informed consent
* Have successfully initiated PrEP and are returning for their second bottle of PrEP pills
* Able to provide a home address or personal telephone number, or able to provide two personal contacts who will be able to know the patient's whereabouts during the study period

Exclusion Criteria

* Under 18 years of age
* Unable to give informed consent due to severe mental or physical illness/substance intoxication at baseline visit
* Presents with severe adverse reactions to PrEP
* The subject will be excluded from the study at his own request for any reason since participation is voluntary

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 310 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
ARV Hair Concentrations | 6 months
  Level of ARV (TDF/FTC) in scalp hair samples

SECONDARY OUTCOMES:
Clinic attendance/retention | 6 months
  This is a measure of retention in care. As each participant finishes his 6-month study period, retention will be determined by number of quarterly care visits completed.
Medication adherence | 6 months
  Medication Possession Ratio (MPR) is defined as the number of dispensed pills divided by the number of days between visits which will be derived from pharmacy refill records
Questionnaire to Assess Self-reported PrEP Use | 6 months
  Self report adherence to assess for change in adherence.
Reduction in HIV and STI incidence relative to control group | 6 months
  Male sex worker participants will be tested at baseline and 6-month follow-up for HIV and syphilis. Incidence rates for all infections at 6-month follow-up will be compared between the conditional economic incentive (CEI) group and the standard of care (SOC) group.
Reduction in number of unprotected sex acts relative to control group | 6 months
  Male sex worker participants will be assessed at baseline and 6-month follow-up using self-report measures of frequency of protected and unprotected sex acts with clients. Changes in frequency at 6-month follow-up will be compared between the conditional economic incentive (CEI) group and the standard of care (SOC) group.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Galarraga, PhD, Principal Investigator — Brown University
Locations (1):
- National Institute of Public Health (INSP) / Clinica Condesa, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Materials generated under this project will be disseminated according to University and NIH policies regarding data sharing. Aggregate-level data collected in this collaboration will ultimately be available for public use. Opportunities for secondary analyses will be available following completion of the three-year project and publication of the main study findings. These findings will be available to the public through scientific meetings and peer-reviewed journals, as well as through a structured policy dissemination process.

REFERENCES:
- [Background] Kadiamada-Ibarra H, Hawley NL, Sosa-Rubi SG, Wilson-Barthes M, Franco RR, Galarraga O. Barriers and facilitators to pre-exposure prophylaxis uptake among male sex workers in Mexico: an application of the RE-AIM framework. BMC Public Health. 2021 Nov 27;21(1):2174. doi: 10.1186/s12889-021-12167-9. PMID 34837988
- [Background] Reichheld SJ, Pellowski JA, Wilson-Barthes M, Galarraga O. Barriers and facilitators to scaling up access to HIV pre-exposure prophylaxis among key populations: A qualitative study of the incentive-based PrEP Seguro program in Mexico. SSM Qual Res Health. 2023 Dec;4:100357. doi: 10.1016/j.ssmqr.2023.100357. Epub 2023 Nov 8. PMID 38099208
- [Result] Salinas-Rodriguez A, Sosa-Rubi SG, Chivardi C, Rodriguez-Franco R, Gandhi M, Mayer KH, Operario D, Gras-Allain N, Vargas-Guadarrama G, Galarraga O. Preferences for Conditional Economic Incentives to Improve Pre-exposure Prophylaxis Adherence: A Discrete Choice Experiment Among Male Sex Workers in Mexico. AIDS Behav. 2022 Mar;26(3):833-842. doi: 10.1007/s10461-021-03443-1. Epub 2021 Aug 27. PMID 34453239
- [Result] Galarraga O, Wilson-Barthes M, Chivardi C, Gras-Allain N, Alarid-Escudero F, Gandhi M, Mayer KH, Operario D. Incentivizing adherence to pre-exposure prophylaxis for HIV prevention: a randomized pilot trial among male sex workers in Mexico. Eur J Health Econ. 2025 Mar;26(2):299-311. doi: 10.1007/s10198-024-01705-y. Epub 2024 Jul 13. PMID 39002005
- [Derived] Chivardi C, Zamudio-Sosa A, Wilson-Barthes M, Alarid-Escudero F, Gandhi M, Mayer KH, Operario D, Galarraga O. Cost-Effectiveness of Using Conditional Economic Incentives to Improve Pre-exposure Prophylaxis Adherence Among Male Sex Workers. Pharmacoecon Open. 2025 Jul;9(4):649-659. doi: 10.1007/s41669-025-00569-z. Epub 2025 Apr 9. PMID 40205318